CLINICAL TRIAL: NCT06727253
Title: GlycanTrigger - WP4: Glycan Supplementation on a Human Model of Crohn's Disease Initiation and Progression: a Pilot Trial
Brief Title: Glycan Supplementation on a Human Model of Crohn's Disease Initiation and Progression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GLSMED Learning Health S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GlycanTrigger
Record Dates: First submitted 2024-11-20; First posted 2024-12-10 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease | interventions — Polysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm, Dietary Supplement: Glycan (Experimental)
  Interventions: Dietary Supplement: Glycan

INTERVENTIONS:
Dietary Supplement: Glycan — The post-operative CD patients will receive an orally administered glycan.

SUMMARY:
The overall aim of this proof-of-concept trial is to investigate the effect of an orally administered glycan on the modulation of the dysregulation of host-microbiome interactions and its effect on the mucosal immune response. Post-operative Crohn's Disease patients will be used as a representative model to mimic the immunopathogenic pathway of health-to-disease transition. Changes in gut glycocalyx seem to be a primary event involved in the disruption of the interaction between the microbiota and the host immune system. Thus, this study aims to assess the effect of the modulation of the glycome on the microbial and immunological changes that contribute to disease development.

DETAILED DESCRIPTION:
Inclusion Criteria

* Male or female patients between 18 and 75 years old able to provide oral and written informed consent for participation in the study
* Confirmed diagnosis of ileal or ileocolonic CD
* Submitted to ICR or ileal resection for removing the diseased segment of the bowel.

Exclusion Criteria

* Diagnosis of indeterminate colitis, ulcerative colitis or microscopic colitis, including collagenous colitis or lymphocytic colitis
* Patients receiving antibiotics, aminosalicylates, thiopurines, methotrexate, biologics or small molecules after surgery for postoperative recurrence
* Patients with previous ICR or ileal resection due to CD, unless the treating physician does not intend to start other prophylactic therapy apart from the glycan supplement within the first 6 months following surgery
* Pregnant or lactating women
* Documented allergy to shellfish, glycans or glycans derivatives
* History of dysplasia on colonic biopsy
* Presence of, or history of cancer, except for skin cancer
* History of poorly controlled type 1 or type 2 diabetes, defined as HbA1c greater than 8% or recurrent episodes of hyperglycaemic crisis such as diabetic ketoacidosis or hyperglycaemic hyperosmolar state
* Patients with known bleeding disorders, such as hemophilia or thrombocytopenia, or those receiving anticoagulation therapy, such as warfarin or direct oral anticoagulants
* Any physical or mental condition which would interfere with the ability to provide written and oral free informed consent or limit the study participation, collection of data, or study completion as determined by the Investigator
* Unwillingness or inability to follow the procedures outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years old (inclusive) able to provide oral and written informed consent for participation in the study
* Confirmed diagnosis of ileal or ileocolonic CD (according to ECCO guidelines)
* Patients submitted to ileal and ileocecal resection for removing the diseased segment of the bowel.

Exclusion Criteria:

* Diagnosis of indeterminate colitis, ulcerative colitis or microscopic colitis (collagenous colitis or lymphocytic colitis)
* Patients receiving antibiotics, aminosalicylates, thiopurines, methotrexate, biologics or small molecules after surgery for postoperative recurrence
* Patients with previous ICR or ileal resection due to CD, unless the treating physician does not intend to start other prophylactic therapy apart from the glycan supplement within the first 6 months following surgery
* Pregnant or lactating women
* Documented allergy to shellfish, glycans or glycans derivatives
* History of dysplasia on colonic biopsy
* Presence of, or history of cancer, except for skin cancer
* History of poorly controlled type 1 or type 2 diabetes (HbA1c>8% or recurrent episodes of hyperglycaemic crisis such as diabetic ketoacidosis or hyperglycaemic hyperosmolar state)
* Patients with known bleeding disorders (e.g. haemophilia or thrombocytopenia) or anticoagulation therapy (e.g. warfarin or direct oral anticoagulants)
* Any physical or mental condition which would interfere with the ability to provide written and oral free informed consent or limit the study participation, collection of data, or study completion as determined by the Investigator
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The effect of the modulation of the glycome on the microbial changes that contribute to disease development | From enrolment until 6 months following surgery
The effect of the modulation of the glycome on the immunological changes that contribute to disease development | From enrolment until 6 months following surgery

SECONDARY OUTCOMES:
The immunomodulatory effect of glycans on endoscopic recurrence | From enrolment until 6 months following surgery
The immunomodulatory effect of glycans on clinical recurrence | From enrolment until 6 months following surgery
The immunomodulatory effect of glycans on histological recurrence | From enrolment until 6 months following surgery
The immunomodulatory effect of glycans on systemic inflammatory biomarkers pre-surgery | From enrolment until 6 months following surgery
The immunomodulatory effect of glycans on systemic inflammatory biomarkers post-surgery | From enrolment until 6 months following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital da Luz Lisboa, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No